CLINICAL TRIAL: NCT06078085
Title: Abdominal Rectus Diastasis Microscopy and Rehabilitation
Brief Title: Abdominal Rectus Diastasis Microscopy and Rehabilitation (AMIRE)
Acronym: AMIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karin Strigård, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-06512-01
Record Dates: First submitted 2023-09-29; First posted 2023-10-11 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Abdominal Rectus Diastasis
Keywords: Randomised controlled trial; Rehabilitation

STUDY DESIGN:
Intervention Model Description: One intervention group that receive a postoperative rehabilitation programme. One control group that can train freely.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 24 patients that receive a postoperative rehabilitation program to follow after they undergo surgery for abdominal rectus diastasis.
  Interventions: Other: Postoperative rehabilitation program
- Control (No Intervention): 24 patients that undergo surgery for abdominal rectus diastasis and can exercise freely after surgery.

INTERVENTIONS:
Other: Postoperative rehabilitation program — The rehabilitation program is created by a physical therapist
  Arms: Intervention

SUMMARY:
The goal of this randomised controlled trial is to evaluate the effect of a postoperative rehabilitation program after surgical correction of abdominal rectus diastasis. The main questions to answer are:

1. Does structured postoperative abdominal exercise improve abdominal wall function in three months and twelve months after surgical correction of abdominal rectus diastasis
2. Does connective tissue components differ in patients with abdominal rectus diastasis when compared to healthy individuals?

DETAILED DESCRIPTION:
The investigators want to include patients in Sweden that are eligible for surgical correction of their abdominal rectus diastasis. Patients will be recruited at the surgical clinic at four hospitals in Sweden. After being informed about the study and potential risks, all patient give written informed consent. Randomisation is performed upon inclusion.

All patients undergo surgery by plication of the linea alba. A blood sample is collected prior to the surgery. During the surgery the skin, connective tissue and rectus muscle are biopsied. On the first postoperative day, another blood sample is collected. Follow up is conducted three and twelve months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diastasis > 3 cm
* At least 1 year since child birth
* One year of steady weight after weightloss
* BMI < 30
* Males with diastasis above and below umbilicus

Exclusion Criteria:

* New planned pregnancy
* Smoker
* Connective tissue disease
* Immunosuppressive treatment
* Umbilical hernia > 2 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
5 times sit to stand test time | Three and twelve months after surgery
  Abdominal wall function measured with the 5 times sit to stand test
Number of repetitions of deadlift with 20 kilograms | Three and twelve months after surgery
  Abdominal wall function measured

SECONDARY OUTCOMES:
VHPQ | Three and twelve months after surgery
  Ventral hernia pain questionnaire collect information on the patients experience of pain
PDI-score | Three and twelve months after surgery
  Pain disability index collect information on how pain influence daily life attributes. Minimum score 0, maximum score 70. A lower score means less disability.
PGPQ | Three and twelve months after surgery
  Patient goal priority questionnaire collect information on activities the patient wish to improve using the intervention
PFDI-20 short form | Three and twelve months after surgery
  Pelvic floor disability index short form collect information on symptoms from the urogenital organs. Minimum score 0, maximum score 40. Absence of symptoms (score 0), symptoms with mild distress (1-15), symptoms with moderate distress (16-34), symptoms with severe distress (35-40).

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Surgical clinic at Mora Hospital, Mora, Dalarna County
  - Surgical clinic at Gällivare Hospital, Gällivare, Norrbotten County
  - Surgical clinic at the district hospital of Skellefteå, Skellefteå, Västerbotten County
  - University Hospital of Umeå, Umeå, Västerbotten County

IPD SHARING:
Plan to Share IPD: Undecided